CLINICAL TRIAL: NCT06996002
Title: Effects of Rhomboids Strength Training Regime on Pain, Craniovertebral Angle and Disability Among Patients With Upper Crossed Syndrome
Brief Title: Effects of Rhomboids Strength Training Regime Among Patients With Upper Crossed Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0145 Bisma
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Upper Crossed Syndrome
Keywords: Craniovertebral Angle; Pain; Disability
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhomboids strengthening exercises along with conventional Exercises (Experimental): Rhomboids strengthening exercises:
  1. Seated Bent Row
  2. Bent Over Row
  3. Lat Pull Down
  4. Shoulder Horizontal Abduction
  5. Band pull apart
  6. Prone lateral raise
  hot pack for 10 min. Trans-cutaneous Electric Nerve Stimulation (TENS). Stretching chest muscles, pectoralis muscles, levator scapulae muscle, cervical extensor muscles, upper trapezius Posture correction exercises
  Interventions: Other: Rhomboids Strengthening Exercise; Other: Conventional Exercises
- Conventional Exercises (Active Comparator): * Both groups will receive hot pack for 10 min.
  * Trans-cutaneous Electric Nerve Stimulation (TENS). Stretching chest muscles, pectoralis muscles, levator scapulae muscle, cervical extensor muscles, upper trapezius
  * Posture correction exercises
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Rhomboids Strengthening Exercise — 1. Seated Bent Row in Sitting position,3 sets of the exercise program with 12 repetitions per set, 3 times per week.
  2. Bent Over Row in standing position, 3 sets, 12 repetitions, 3 times per week.
  3. Lat Pull Down in sitting position with 12 repetitions per set, 3 times per week.
  4. Shoulder Horizontal Abduction in lying position with 3 sets of the exercise program with 12 repetitions per set, 3 times per week.
  5. Band pull apart performed 4sets, 12 repetitions, and 10 seconds rest for 2 mints, 3 times per week.
  6. Prone lateral raise with 3 sets of the exercise program with 12 repetitions per set, 3 times per week.
  Conventional treatment Modalities:
  Trans-cutaneous Electric Nerve Stimulation (TENS) and Hot pack, postural exercises and stretching exercises
  Arms: Rhomboids strengthening exercises along with conventional Exercises
Other: Conventional Exercises — Conventional Treatment
  1. hot pack for 10 min,
  2. Trans-cutaneous Electric Nerve Stimulation (TENS) will be applied, with pulse duration of 250 microseconds at a frequency of 80 Hz for 15 min in the sub occipital region and the trapezius bilaterally.
  3. Stretching exercises of tight muscles 2 sets of 15 min.
  4. Posture correction exercises:
  releasing muscles of anterior part of the trunk, neck, shoulder.

SUMMARY:
Upper Cross Syndrome (UCS) is characterized by weakening of the neck flexors and rhomboids and stiffness in the pectoralis major, upper trapezius, and levator scapulae. Rhomboids major and minor need to be strengthened in order to enhance scapular stability and regain proper posture. The aim of this study is to determine effect of rhomboids strength training regime on pain, craniovertebral angle and disability among patients with upper crossed syndrome.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Haleema Surgical Hospital, Shorkot city. Non-probability convenient sampling will be used to collect the data. Sample size of 38 subjects with age group between 20-45 years will be taken. Data will be collected from the patients having present complaint of upper crossed syndrome pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, craniovertebral angle, and neck disability index questionnaire for disability. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by computer-generated stratified randomization. The study will be a single-blind assessor. Both the Groups will receive Hot Pack, TENS, posture training and stretching exercises while group A will receive rhomboids strengthening exercises additionally. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 20 and 45 years
* Both gender male and female
* Subject with head neck angle less than 50 degrees(for forward head posture).
* Subject with positive JANDAS upper crossed syndrome tests .
* Population with occupation tailor, computer users and students.

Exclusion Criteria:

* • Exclusion criteria Patients were excluded if they were diagnosed with the following conditions for ˃6 months

  * Tuberculosis, carcinoma, heart disease, and osteoporosis
  * Neural disorders due to prolapsed intervertebral disc
  * Any trauma or localized infection in upper back region

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10.
  0 indicates "no pain" 1-3 indicate "Mild pain" 4-6 indicate "Moderate pain" 7-10 indicate "worst pain". NPRS have shown high test-retest reliability (r = 0.96 and 0.95, respectively)
Neck Disability Index (NDI_ | upto 4 weeks
  The NDI is a 10-item, 50-point index that evaluates many facets of day-to-day functioning in individuals with neck pain. The NDI evaluates two items pertaining to discretionary daily living activities (personal care, reading), four items pertaining to activities of daily living (lifting, work, driving, and recreation), and four items related subjective symptoms (pain intensity, headache, concentration, and sleeping). The scores are interpreted as follows:
  0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability 35-50: Complete disability. For the NDI, test-retest reliability was good
Craniovertebral Angle | upto 4 weeks
  Anatomically speaking, the degree of forward head posture is measured using the craniovertebral angle (CVA), which is a measurement of the head and neck posture. It is the angle created by a horizontal line running from the C7 vertebra and the line joining the tragus of the ear to the vertebra (the seventh cervical vertebra).
  In order to calculate the craniovertebral angle:
  1. Indicate the C7 vertebra and the tragus of the ear.
  2. Draw an imaginary line that connects the C7 vertebra to the tragus.
  3. Sketch a line that extends horizontally from the vertebra C7.
  4. Calculate the angle that these two lines form. More than 50 degrees is the normal CVA. Head tilt slightly forward, between 40 and 50 degrees. A somewhat forward head posture, between 30 and 40 degrees. Head Posture Severe Forward when it is less than 30 degrees. CVA is a trustworthy measure of head and neck posture

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD Scholar, Principal Investigator — Riphah International University
Locations (1):
- Haleema Surgical Hospital, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mujawar JC, Sagar JH. Prevalence of Upper Cross Syndrome in Laundry Workers. Indian J Occup Environ Med. 2019 Jan-Apr;23(1):54-56. doi: 10.4103/ijoem.IJOEM_169_18. PMID 31040591
- [Background] Jeong GH, Lee BH. Effects of Telerehabilitation Combining Diaphragmatic Breathing Re-Education and Shoulder Stabilization Exercises on Neck Pain, Posture, and Function in Young Adult Men with Upper Crossed Syndrome: A Randomized Controlled Trial. J Clin Med. 2024 Mar 11;13(6):1612. doi: 10.3390/jcm13061612. PMID 38541838
- [Background] Naseer R, Tauqeer S. Prevalence of upper cross syndrome in different occupations. Pakistan Journal of Physical Therapy (PJPT). 2021:03-7.
- [Background] Huang JF, Meng Z, Zheng XQ, Qin Z, Sun XL, Zhang K, Tian HJ, Wang XB, Gao Z, Li YM, Wu AM. Real-World Evidence in Prescription Medication Use Among U.S. Adults with Neck Pain. Pain Ther. 2020 Dec;9(2):637-655. doi: 10.1007/s40122-020-00193-1. Epub 2020 Sep 17. PMID 32940899
- [Background] Chu EC, Butler KR. Resolution of Gastroesophageal Reflux Disease Following Correction for Upper Cross Syndrome-A Case Study and Brief Review. Clin Pract. 2021 May 21;11(2):322-326. doi: 10.3390/clinpract11020045. PMID 34063944
- [Background] Kirthika SV, Sudhakar S, Padmanabhan K, Ramanathan K. Impact of upper crossed syndrome on pulmonary function among the recreational male players: A preliminary report. Saudi Journal of Sports Medicine. 2018;18(2):71-4.
- [Background] Gull M, Akbar UU, Asim HM. FREQUENCY OF CHRONIC NECK PAIN IN UPPER CROSS SYNDROME IN FEMALE SCHOOL TEACHERS. Independent Journal of Allied Health Sciences. 2018;1(01):33-8.
- [Background] Firouzjah MH, Firouzjah EMAN, Ebrahimi Z. The effect of a course of selected corrective exercises on posture, scapula-humeral rhythm and performance of adolescent volleyball players with upper cross syndrome. BMC Musculoskelet Disord. 2023 Jun 14;24(1):489. doi: 10.1186/s12891-023-06592-7. PMID 37316911